CLINICAL TRIAL: NCT05409859
Title: Assessing Adverse Events Associated With Manual Therapies in Preschool Pediatric Population: a Feasibility Study
Brief Title: Adverse Events Associated With Manual Therapies in Children
Status: Completed | Type: Observational
Sponsor: Université du Québec à Trois-Rivières (Other)
Responsible Party: Sponsor
Other Study IDs: UQTR_peds_2021-2022
Record Dates: First submitted 2022-06-03; First posted 2022-06-08 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Adverse Event
Keywords: Manual therapy; Spinal mobilization; Complementary and alternative therapy; Pediatric; Chiropractic
MeSH Terms: interventions — Musculoskeletal Manipulations; Therapy, Soft Tissue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Children patients of 5 years and younger who received manual therapies by a chiropractor in private practice.
  Interventions: Other: Manual therapies

INTERVENTIONS:
Other: Manual therapies — Manual therapies were determined based on the clinician evaluation and could include spinal mobilization delivered by hands or mechanically assisted and soft tissue therapies.
  Other Names: Manual therapy; Spinal mobilization delivered by hands; Soft tissue therapy; Mechanically assisted spinal mobilization

SUMMARY:
This study aims to evaluate the feasibility to conduct a prospective cohort study evaluating the adverse events associated with manual therapies in children of 5 years and younger. A validated reporting system will be used to evaluate the adverse events and include a total of four questionnaires that are filled online. Adverse events will be evaluated immediately following the intervention and at 48h post-intervention.

DETAILED DESCRIPTION:
The aim of this study is to investigate (1) the feasibility to conduct a prospective cohort study evaluating the adverse events associated with manual therapies in children of 5 years and younger and (2) to report preliminary data on the frequency and nature of the adverse events. Participating chiropractors will advertise the study in their private clinic through flyers and posters. Legal tutors interested to participate will access an information sheet and consent form using a link available on the flyers/posters. Legal tutors of participants will complete three questionnaires, one before the intervention to describe the child (e.g. age, sex, reason(s) to seek care), one immediately following the intervention to report immediate adverse events and one 48h following the intervention to report delayed adverse events. Clinicians will complete one questionnaire immediately following the intervention to describe the manual therapies delivered to the children. All questionnaires will be available online on a secured platform. The intervention will be determined by the clinician according the their evaluation of the child and could include spinal mobilization as well as soft tissue therapies.

ELIGIBILITY:
Inclusion Criteria:

* Children of 5 years or younger
* First or second treatment at one of the chiropractic clinic
* Spinal mobilization has to be clinically indicated

Exclusion Criteria:

* Children of 6 years or older
* Spinal mobilization not indicated

Max Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children of 5 years or less consulting at one of the participating chiropractors' private practice localized in Québec province (Canada).
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Immediate adverse event | 5 minutes following the intervention
  New symptom or aggravation of a preexisting symptom noted by the legal tutor of the children immediately following the manual therapies
Delayed adverse event | 48 hours following the intervention
  New symptom or aggravation of a preexisting symptom noted by the legal tutor of the children 48h following the manual therapies

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Pagé, PhD, Principal Investigator — Université du Québec à Trois-Rivières
Locations (1):
- Université du Québec à Trois-Rivières, Trois-Rivières, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dolbec A, Doucet C, Pohlman KA, Sobczak S, Page I. Assessing adverse events associated with chiropractic care in preschool pediatric population: a feasibility study. Chiropr Man Therap. 2024 Mar 13;32(1):9. doi: 10.1186/s12998-024-00529-0. PMID 38481318